CLINICAL TRIAL: NCT06848712
Title: Brain Structural Abnormalities in Patients With Vertigo
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: IG/296-1/2025/2
Record Dates: First submitted 2025-02-11; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Vertigo; MRI
Keywords: vertigo; MRI; white matter lesions; Circle of Willis; sinusitis; BPPV; lifestyle modifications; betahistine
MeSH Terms: conditions — Vertigo; Sinusitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Vertigo Group: Participants in this group reported dizziness as a primary symptom and were referred for brain MRI to investigate potential structural abnormalities. Exclusion criteria included any pre-existing neurological disorders. The most common diagnoses after MRI included benign paroxysmal positional vertigo (BPPV) and vertebrobasilar syndrome.
  Interventions: Other: Observational Study - No intervention
- Control Group: Participants in this group did not report dizziness or other neurological symptoms. They underwent brain MRI for other reasons but had no history of neurological disorders. This group served as a comparison to evaluate the prevalence of brain structural abnormalities in vertigo patients.
  Interventions: Other: Observational Study - No intervention

INTERVENTIONS:
Other: Observational Study - No intervention — This is an observational study evaluating brain structural abnormalities in post-COVID headache patients. No experimental intervention is applied.

SUMMARY:
Introduction: Dizziness is one of the most common complaints in medical practice and is associated with various underlying conditions, including neurological, otolaryngological, and psychological disorders. Preliminary imaging studies like CT, cervical spine X-rays, and carotid/vertebral artery ultrasound, aids in precise diagnosis and targeted therapeutic decisions. MRI is one of the most effective imaging modalities currently available for examining the brain.

Purpose: To identify structural brain changes linked to vertigo, explore pre-MRI diagnostic approaches, and evaluate treatment strategies.

Methods: The study included 232 patients with vertigo and 232 control subjects. MRI results were categorized, and pre-MRI examinations, symptoms, and treatments were analyzed. Statistical comparisons were conducted using chi-square and t-tests, with significance set at p<0.05.

DETAILED DESCRIPTION:
Vertigo is a prevalent symptom with multiple underlying etiologies, including neurological, vascular, and musculoskeletal causes. Despite its high prevalence, the exact structural brain abnormalities associated with vertigo remain unclear. This observational study aims to assess brain MRI findings in patients with vertigo and compare them to a control group without vertigo symptoms. The study also evaluates pre-MRI diagnostic procedures, such as vertebral/carotid ultrasound and cervical spine X-rays, to identify potential vascular and musculoskeletal contributors to vertigo. The results may provide insights into the structural brain changes linked to vertigo and help refine diagnostic and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Reported dizziness (vertigo) as a primary symptom
* Brain MRI requested by the attending physician

Exclusion Criteria:

* Prior neurological disease or disorder (other than vertigo/dizziness in the vertigo group)
* MRI contraindications (e.g., pacemaker, metal implants, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients (≥18 years) with vertigo who were referred for brain MRI to investigate potential structural abnormalities. A control group of individuals without a history of vertigo or neurological disorders was included for comparison. Exclusion criteria included prior neurological diseases, recent head trauma, and MRI contraindications.
Sampling Method: Non-Probability Sample
Enrollment: 464 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrences With Specific Structural Brain Abnormalities Observed on MRI | From September 2020 to December 2022
  Brain MRI findings were analyzed to compare the occurrences of structural abnormalities between vertigo patients and control participants. The most commonly assessed abnormalities included white matter lesions, lacunar infarcts, Circle of Willis variations, and sinusitis. The occurrences (number and percentage) of these findings in each group will be compared using chi-square tests.

SECONDARY OUTCOMES:
Occurrences of associated symptoms in vertigo patients | From September 2020 to December 2022
  The study evaluated the occurrences of associated symptoms, including headache, imbalance, visual disturbances, and psychological symptoms (anxiety and depression). Each symptom's occurrences (number and percentage) will be reported separately.
Occurrences of pre-MRI diagnostic procedures in vertigo patients | From September 2020 to December 2022
  The study assessed the occurrences of patients with vertigo undergoing pre-MRI diagnostic procedures, including carotid/vertebral ultrasound and cervical spine X-rays. Each procedure's occurrences (number and percentage) will be reported separately.
Occurrences of post-MRI diagnoses in vertigo patients | From September 2020 to December 2022
  The study analyzed the most common diagnoses after MRI, including vestibular migraine, benign paroxysmal positional vertigo (BPPV), and vascular dizziness. Each diagnosis's occurrences (number and percentage) will be reported separately.
Occurrences of treatment strategies applied | From September 2020 to December 2022
  The study evaluated the most frequent treatment strategies, including physical therapy, pharmacological treatment (e.g., betahistine), and lifestyle modifications. Each treatment's occurrences (number and percentage) will be reported separately.

CONTACTS AND LOCATIONS:
Overall Officials: Klaudia Széphelyi, Principal Investigator — University of Pécs, Faculty of Health Sciences, Hungary
Locations (1):
- Szent Margit Hospital, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szephelyi K, Kora S, Orsi G, Tollar J. Structural Brain Abnormalities, Diagnostic Approaches, and Treatment Strategies in Vertigo: A Case-Control Study. Neurol Int. 2025 Sep 10;17(9):146. doi: 10.3390/neurolint17090146. PMID 41002934